CLINICAL TRIAL: NCT03270384
Title: Re-establishing Flow Via Drug Coated Balloon For The Treatment Of Urethral Stricture Disease
Acronym: ROBUST-II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Urotronic Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: PR1032
Record Dates: First submitted 2017-08-30; First posted 2017-09-01 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-07

CONDITIONS: Urethral Stricture
Keywords: early feasibility; non-randomized
MeSH Terms: conditions — Urethral Stricture

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Treatment (Experimental): Up to 15 subjects will be enrolled and treated with the Urotronic drug coated balloon (DCB)
  Interventions: Device: Urotronic Drug Coated Balloon (DCB)

INTERVENTIONS:
Device: Urotronic Drug Coated Balloon (DCB) — The Urotronic Drug Coated Balloon (DCB) is a guidewire compatible catheter with a tapered atraumatic tip. The distal end of the catheter has an inflatable balloon coated with a proprietary coating containing the drug paclitaxel that facilitates the drug's transfer to the urethral wall upon inflation.

SUMMARY:
The study described below is designed to assess the safety and device performance for the drug coated balloon (DCB) for the treatment of urethral stricture.

ELIGIBILITY:
Inclusion Criteria:

1. Male subjects ≥ 18 years' old
2. Visual confirmation of stricture via cystoscopy or urethrogram
3. Single lesion anterior urethral stricture less than or equal to 3 cm
4. Two (2) or more prior diagnosis and treatment of stricture treatments (including self-catheterization) including DVIU (direct visual internal urethrotomy), but no prior urethroplasty
5. Significant symptoms of stricture such as frequency of urination, dysuria, urgency, hematuria, slow flow, feeling of incomplete emptying, recurrent UTI's (urinary tract infections).
6. IPSS (International Prostate Symptom Score) score of 13 or higher
7. Lumen diameter <12F by urethrogram
8. Able to complete validated questionnaire independently
9. Qmax <12 ml/sec
10. Guidewire must be able to cross the lesion

Exclusion Criteria:

1. Strictures greater than 3.0 cm long.
2. Subjects that have more than 1 stricture.
3. Sensitivity to paclitaxel or on medication that may have negative interaction with paclitaxel
4. Subjects who have a suprapubic catheter
5. Previous urethroplasty within the anterior urethra
6. Stricture due to bacterial urethritis or untreated gonorrhea
7. Stricture dilated or incised within the last 3 months
8. History of over active bladder or stress incontinence
9. Previous radical prostatectomy
10. Previous pelvic radiation
11. Diagnosed kidney, bladder, urethral or ureteral stones or active stone passage in the past 6 months.
12. Presence of a penile implant, artificial urinary sphincter, or stent(s) in the urethra or prostate
13. Known neurogenic bladder, sphincter abnormalities, or poor detrusor muscle function

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2017-10-25 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2025-02-19 (Actual)

PRIMARY OUTCOMES:
Safety- Rate of Device Related Serious Complications | 90 days

SECONDARY OUTCOMES:
Safety- Change in IIEF (International Index of Erectile Function) | 90 days
Efficacy- Stricture Recurrence Rate | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Sean Elliott, MD, Principal Investigator — University of Minnesota
Locations (5):
- United States (5):
  - University of Iowa, Iowa City, Iowa
  - Chesapeake Urology, Hanover, Maryland
  - University of Minnesota, Minneapolis, Minnesota
  - Metro Urology, Woodbury, Minnesota
  - Urology of Virginia, Virginia Beach, Virginia

IPD SHARING:
Plan to Share IPD: Undecided